CLINICAL TRIAL: NCT01274897
Title: A Phase 3, Multi-center, Observer-blind, Placebo-controlled, Randomized Study to Evaluate the Immunogenicity and Safety of Novartis Meningococcal ACWY Conjugate Vaccine in Healthy Subjects From 11 to 55 Years of Age in Korea
Brief Title: A Multi-center, Observer-blind, Placebo-controlled, Randomized Study to Evaluate the Immunogenicity and Safety of MenACWY in Adolescents and Adults in Korea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V59_39
Record Dates: First submitted 2011-01-09; First posted 2011-01-12 (Estimated); Results first posted 2012-10-16 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-09

CONDITIONS: Meningococcal Disease; Meningococcal Meningitis
Keywords: Meningococcal; ACWY-CRM; Conjugate Vaccine; Meningitis; Adolescents; Persistence; Adults
MeSH Terms: conditions — Meningococcal Infections; Meningitis, Meningococcal; Meningitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MenACWY-CRM (Experimental): Subjects received one dose of MenACWY-CRM conjugate vaccine.
  Interventions: Biological: Novartis MenACWY-CRM
- Placebo (Placebo Comparator): Subjects received the saline placebo.
  Interventions: Biological: Saline Placebo

INTERVENTIONS:
Biological: Novartis MenACWY-CRM — All subjects had blood drawn at Day 1 and Day 29.
  Arms: MenACWY-CRM
Biological: Saline Placebo — All subjects had blood drawn at Day 1 and Day 29.
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the immunogenicity and the safety of a quadrivalent vaccine MenACWY-CRM in healthy subjects from 11 to 55 years of age in Korea.

ELIGIBILITY:
Inclusion Criteria:

Individuals eligible for enrollment in this study were those:

1. who were 11-55 years of age inclusive and who, after the nature of the study had been explained:

   1. had given written assent and/or for whom the parent/legal representative had provided written informed consent (11-19 years of age).
   2. had provided written informed consent (20-55 years of age).
2. who the investigator believed that they or their parents/legal representatives would comply with the requirements of the protocol (e.g., completion of the Diary Card, return for follow-up visit).
3. who were in good health as determined by

   1. medical history
   2. physical assessment
   3. clinical judgment of the investigator
4. who had negative urine pregnancy test for women of childbearing age.

Exclusion Criteria:

Individuals not eligible to be enrolled in the study were those:

1. who were unwilling or unable to give written informed assent or consent to participate in the study.
2. who were perceived to be unreliable or unavailable for the duration of the study period.
3. who were planning to leave the area of the study site before the end of the study period.
4. who had a previous or suspected disease caused by N. meningitidis.
5. who had household contact with and/or intimate exposure to an individual with culture-proven N. meningitidis infection within 60 days prior to enrollment.
6. who had previously been immunized with a meningococcal vaccine.
7. who had received any investigational or non-registered product (drug or vaccine)within 28 days prior to enrollment or who expected to receive an investigational drug or vaccine prior to the completion of the study.
8. who had received any licensed vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrollment in this study or who were planning to receive any vaccine within 30 days from the study vaccines. (Exception: Influenza vaccine was administered up to 15 days prior to study vaccination and at least 15 days after study vaccination)
9. who had experienced within the 7 days prior to enrollment significant acute or chronic infection (for example requiring systemic antibiotic treatment or antiviral therapy) or had experienced fever (defined as body temperature ≥38°C) within 3 days prior to enrollment.
10. who had any serious acute, chronic or progressive disease (e.g., any history of neoplasm, cancer, diabetes, cardiac disease, autoimmune disease, HIV infection or AIDS, or blood dyscrasias, with signs of cardiac or renal failure or severe malnutrition).
11. who had epilepsy or any progressive neurological disease.
12. who had a history of any anaphylaxis, serious vaccine reactions, or allergy to any vaccine components, including latex allergies.
13. who had a known or suspected impairment/alteration of immune function, either congenital or acquired or resulting from (for example):

    1. received immunosuppressive therapy within 28 days prior to enrollment(any systemic corticosteroid administered for more than 5 days, or in a daily dose > 1 mg/kg/day prednisone or equivalent during any of 28 days prior to enrollment, or cancer chemotherapy)
    2. received immunostimulants
    3. received parenteral immunoglobulin preparation, blood products, and/or plasma derivatives within 90 days prior to enrollment and for the full length of the study
14. who were known to have a bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.
15. who had any condition that, in the opinion of the investigator, might interfere with the evaluation of the study objectives.

Ages: 11 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 450 (Actual)
Dates: Start 2010-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines and Diagnostics, Study Chair — Novartis Vaccines
Locations (8):
- South Korea (8):
  - Department of Pediatrics, Kosin University Gospel Hospital, Busan
  - Department of Pediatrics, Seoul National University Bundang Hospital, Gyeonggi-do
  - Deaprtment of Pediatrics, Inha University Hospital, Incheon
  - Division of Infectious Diseases, Inha University Hospital, Incheon
  - Pediatrics and Adolescent medicine, Myongji Hospital Kwandong University, Kyunggi
  - Department of Pediatrics, Ewha Womans University Mokdong Hospital, Seoul
  - Division of Infection Diseases, Seoul National University Hospital, Seoul
  - Division of Infectious Diseases, Korea University Guro Hospital, Seoul

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 8 centres in the Korea.
Pre-assignment Details: All enrolled subjects were included in the trial.
Period: Overall Study
Arm/Group | MenACWY-CRM | Placebo
Started | 297 | 153
Completed | 297 | 153
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MenACWY-CRM | Placebo | Total
Number analyzed (Participants) | 297 | 153 | 450
Age Continuous [Mean (Standard Deviation); unit: years]
  Age, Years | 19.6 (9.2) | 19.3 (8.9) | 19.5 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 139 | 77 | 216
  Male | 158 | 76 | 234

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Subjects With Seroresponse, Directed Against Neisseria Meningitidis Serogroups A, C, W and Y After MenACWY-CRM Vaccination.
Description: Immunogenicity was measured as the percentage of subjects with hSBA response and associated 95% Clopper-Pearson confidence interval (CI), directed against N. meningitidis serogroups A, C, W and Y by serum bactericidal assay using human complement, human serum bactericidal assay (hSBA), at day 29 (28 days after MenACWY-CRM vaccination).
  Seroresponse is defined as:
  1. for subjects with a pre-vaccination hSBA titer < 1:4, a postvaccination hSBA titer ≥ 1:8.
  2. for subjects with a pre-vaccination hSBA titer ≥ 1:4, an increase in hSBA titer of at least four times the pre-vaccination titer.
Time Frame: day 29
Population: Analysis was done on per protocol (PP) population i.e. the subjects who received the vaccine correctly and provided evaluable serum samples at the relevant time points.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY-CRM | Placebo
Number analyzed (Participants) | 296 | 152
Percentages of subjects
  Serogroup A (N=295,152) | 76 [71 to 81] | 1 [0 to 5]
  Serogroup C (N=293,150) | 86 [82 to 90] | 1 [0 to 5]
  Serogroup W (N=293,151) | 28 [23 to 33] | 4 [1 to 8]
  Serogroup Y (N=294,152) | 69 [63 to 74] | 2 [0 to 6]
Statistical Analysis 1: Comparison: MenACWY-CRM; The null hypothesis associated with the primary immunogenicity objective is that for at least one of the four serogroups, the percentage of subjects with hSBA seroresponse at 29 days postvaccination is < 50%; Test type: Superiority or Other; Clopper and Pearson — The immune response considered sufficient if for serogroup A the lower limit of the two-sided 95% Clopper-Pearson confidence interval (CI) of the percentage of subjects with hSBA seroresponse is ≥50%; Lower limit of the two-sided 95% CI = 71, 95% CI 2-sided [71 to 81] — For serogroup A
Statistical Analysis 2: Comparison: MenACWY-CRM; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Clopper and Pearson — The immune response was considered sufficient if for serogroup C, the lower limit of the two-sided 95% CI of the percentage of subjects with hSBA seroresponse was ≥50%; Lower limit of the two-sided 95% CI = 82, 95% CI 2-sided [82 to 90] — For the serogroup C
Statistical Analysis 3: Comparison: MenACWY-CRM; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Clopper and Pearson — The immune response was considered sufficient if for serogroup W, the lower limit of the two-sided 95% CI of the percentage of subjects with hSBA seroresponse was ≥50%; Lower limit of the two-sided 95% CI = 23, 95% CI 2-sided [23 to 33] — For the serogroup W
Statistical Analysis 4: Comparison: MenACWY-CRM; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Clopper and Pearson — The immune response was considered sufficient if for serogroup Y, the lower limit of the two-sided 95% CI of the percentage of subjects with hSBA seroresponse was ≥50%; Lower limit of the two-sided 95% CI = 63, 95% CI 2-sided [63 to 74] — For serogroup Y

2. Secondary Outcome: Geometric Mean Titers (GMTs) of Subjects, Directed Against N. Meningitidis Serogroups A, C, W and Y After MenACWY-CRM Vaccination.
Description: Immunogenicity was assessed as hSBA GMTs and associated 95% CI, measured against N. meningitidis serogroups A, C, W and Y, before the vaccination (baseline, day 1) and at day 29 (28 days after MenACWY-CRM vaccination).
Time Frame: day 1 and day 29
Population: Analysis was done on PP population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenACWY-CRM | Placebo
Number analyzed (Participants) | 296 | 152
Titers
  Serogroup A at Day 1 (N=295,152) | 2.7 [2.47 to 2.95] | 2.86 [2.53 to 3.24]
  Serogroup A at Day 29 (N=295,152) | 48 [39 to 57] | 3 [2.31 to 3.88]
  Serogroup C at Day 1 (N=293,150) | 7.82 [6.76 to 9.05] | 5.94 [4.85 to 7.27]
  Serogroup C at Day 29 (N=293,150) | 231 [198 to 269] | 6.04 [4.89 to 7.47]
  Serogroup W at Day 1 (N=293,151) | 51 [44 to 61] | 48 [38 to 60]
  Serogroup W at Day 29 (N=293,151) | 147 [125 to 171] | 47 [38 to 58]
  Serogroup Y at Day 1 (N=294,152) | 9.01 [7.64 to 11] | 8.82 [7.02 to 11]
  Serogroup Y at Day 29 (N=294,152) | 107 [89 to 128] | 8.4 [6.54 to 11]

3. Secondary Outcome: Percentages of Subjects With hSBA Titer ≥1:8, Directed Against N. Meningitidis Serogroups A, C, W and Y After MenACWY-CRM Vaccination.
Description: Immunogenicity was measured as the percentage of subjects with hSBA titer ≥1:8 and associated 95% CI, at baseline before vaccination (day 1) and at day 29 (28 days after MenACWY-CRM vaccination).
Time Frame: day 1 and day 29
Population: Analysis was done on PP population.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY-CRM | Placebo
Number analyzed (Participants) | 296 | 152
Percentages of subjects
  Serogroup A at Day 1 (N=295,152) | 13 [9 to 17] | 15 [10 to 22]
  Serogroup A at Day 29 (N=295,152) | 79 [74 to 84] | 16 [10 to 23]
  Serogroup C at Day 1 (N=293,150) | 49 [44 to 55] | 39 [31 to 47]
  Serogroup C at Day 29 (N=293,150) | 99 [97 to 100] | 37 [30 to 46]
  Serogroup W at Day 1 (N=293,151) | 89 [85 to 92] | 87 [80 to 92]
  Serogroup W at Day 29 (N=293,151) | 98 [96 to 99] | 88 [82 to 93]
  Serogroup Y at Day 1 (N=294,152) | 54 [48 to 60] | 53 [44 to 61]
  Serogroup Y at Day 29 (N=294,152) | 94 [91 to 97] | 51 [42 to 59]

4. Secondary Outcome: Number of Subjects Who Reported Local and Systemic Reactogenicity During 7 Days After MenACWY-CRM Vaccination
Time Frame: during 7 days of vaccination
Population: Analysis was done on safety population i.e. the subjects in the exposed population who provided post-baseline safety data.
Measure: Number; unit: Subjects
Arm/Group | MenACWY-CRM | Placebo
Number analyzed (Participants) | 297 | 153
Subjects
  Injection site pain | 69 | 12
  Injection site erythema | 30 | 3
  Injection site induration | 30 | 0
  Chills | 17 | 7
  Nausea | 22 | 10
  Myalgia | 45 | 13
  Arthralgia | 6 | 4
  Headache | 39 | 25
  Rash | 1 | 0
  Fever (≥38°C) | 3 | 1
  Axillary temperature (<38.0°C) | 294 | 152
  Stayed home | 9 | 2
  Used analgesic or antipyretic medicines | 7 | 3

ADVERSE EVENTS:
Time Frame: Throughout the study period (29 days)
Arm/Group | MenACWY-CRM | Placebo
Serious Adverse Events (participants affected / at risk) | 0/297 | 0/153
Other Adverse Events (participants affected / at risk) | 117/297 | 50/153
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MenACWY-CRM (N=297) | Placebo (N=153)
Nausea (Gastrointestinal disorders) | 22 (22) | 10 (10)
Chills (General disorders) | 17 (17) | 7 (7)
Injection site erythema (General disorders) | 30 (30) | 3 (3)
Injection site induration (General disorders) | 30 (30) | 0 (0)
Injection site pain (General disorders) | 69 (69) | 12 (12)
Malaise (General disorders) | 21 (21) | 9 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 46 (46) | 13 (13)
Headache (Nervous system disorders) | 39 (39) | 25 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days